CLINICAL TRIAL: NCT01750151
Title: The Effect of Sedentary Video Game Playing Before a Mixed Meal on Subjective Appetite and Satiety Signals From a Glucose Preload in Normal Weight and Overweight/Obese Boys
Brief Title: Video Game Playing on Lunch-time Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Danone Institute International (Other); Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assistant Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2012-120-001
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Exogenous Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Glucose beverage (Experimental): Glucose beverage
  Interventions: Dietary Supplement: Glucose Beverage
- Control beverage and video game playing (Experimental): Control beverage and video game playing
  Interventions: Behavioral: Video Game Playing
- Glucose beverage and video game playing (Experimental): Glucose beverage and video game playing
  Interventions: Behavioral: Video Game Playing
- Control beverage (Experimental): Control beverage
  Interventions: Dietary Supplement: Control Beverage

INTERVENTIONS:
Dietary Supplement: Glucose Beverage
  Arms: Glucose beverage
Behavioral: Video Game Playing
  Arms: Control beverage and video game playing; Glucose beverage and video game playing
Dietary Supplement: Control Beverage
  Arms: Control beverage

SUMMARY:
The purpose of this experiment is to investigate the effect of video game playing for 30 minutes on food intake and subjective appetite. The investigators hypothesize that video game playing will affect food intake in children. Food intake will be measured at 30 minutes following a glucose (50g glucose in 250ml of water) or sweetened non-caloric (150mg Sucralose® in 250ml of water) beverage with or without video game playing. Subjective appetite will be measured at 0, 20, 35 and 65 minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy boys with no emotional, behavioral or learning problems

Exclusion Criteria:

* girls

Ages: 9 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Food Intake (kcal) | at 30 min after the treatment

SECONDARY OUTCOMES:
Subjective appetite (mm) | 0-65 min
  Subjective appetite (in mm) determined by visual analogue scale will be determined at 0, 20, 35 and 65 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (2):
- Canada (2):
  - Department of Applied Human Nutrition, Halifax, Nova Scotia
  - School of Nutrition, Ryerson University, Toronto, Ontario

REFERENCES:
- [Derived] Branton A, Akhavan T, Gladanac B, Pollard D, Welch J, Rossiter M, Bellissimo N. Pre-meal video game playing and a glucose preload suppress food intake in normal weight boys. Appetite. 2014 Dec;83:256-262. doi: 10.1016/j.appet.2014.08.024. Epub 2014 Aug 20. PMID 25150911